CLINICAL TRIAL: NCT05792865
Title: A Registry Study of Patients Hospitalized With Confirmed COVID-19
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Zhang Yi, professer, Beijing Chao Yang Hospital
Other Study IDs: CYH-PHARM1
Record Dates: First submitted 2023-03-28; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
Keywords: Hospitalized; paxlovid
MeSH Terms: conditions — COVID-19 | interventions — nirmatrelvir and ritonavir drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Biospecimen Retention: Samples Without DNA — Residual specimen, plasma, 1 ml. Each specimen will be uniquely identified to ensure that patient privacy is not compromised.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Paxlovid（Within 5 days after the diagnosis of COVID-19）: According to the patient's medical records, the time from the diagnosis of COVID-19 to the prescription of PAXLOVID is within 5 days.
  Interventions: Drug: paxlovid
- Paxlovid （More than 5 days after the diagnosis of COVID-19）: According to the patient's medical records, the time from the diagnosis of COVID-19 to the prescription of PAXLOVID exceeds 5 days.
  Interventions: Drug: Paxlovid
- No paxlovid used: Patients have never used Paxlovid after being diagnosed with COVID-19, whether before or after hospitalization.
  Interventions: Drug: No paxlovid

INTERVENTIONS:
Drug: paxlovid — Patients treated with PAXLOVID within 5 days of being diagnosed with covid-19 will be included in this group. Patients treated with PAXLOVID will be included in this group. This study is a non-interventional observational study, and no intervention measures were applied to the clinical diagnosis and treatment process of hospitalized COVID-19 patients. The use of Paxlovid is completely decided by the clinical doctors based on the patients' condition and clinical experience.
  Other Names: paxlovid within initial 5 days
  Groups: Paxlovid（Within 5 days after the diagnosis of COVID-19）
Drug: No paxlovid — Patients not treated with PAXLOVID will be included in this group. This study is a non-interventional observational study, and no intervention measures were applied to the clinical diagnosis and treatment process of hospitalized COVID-19 patients. The use of Paxlovid is completely decided by the clinical doctors based on the patients' condition and clinical experience.
  Groups: No paxlovid used
Drug: Paxlovid — Patients treated with PAXLOVID outside of the initial 5 days after being diagnosed with covid-19 will be included in this group.
  Other Names: Paxlovid outside of the initial 5 days
  Groups: Paxlovid （More than 5 days after the diagnosis of COVID-19）

SUMMARY:
The design of this registered study aims to evaluate the efficacy and safety of Paxlovid in the treatment of hospitalized COVID-19 patients, and to explore factors related to the efficacy and safety of Paxlovid.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of COVID-19 infection.
2. Presence of at least one high-risk factor, including age ≥60 years, diabetes, hypertension, cardiovascular disease, stroke, chronic liver or kidney disease, cancer, history of smoking or obesity.

Exclusion Criteria:

* No specific exclusion criteria in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will focus on COVID-19 infected patients who are admitted to the Beijing Chaoyang Hospital, affiliated with Capital Medical University, from November 15th, 2022 to March 30th, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 488 (Estimated)
Dates: Start 2023-03-30 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Disease progression rates | up to 28 days
  The proportion of patients who experienced any of the following events within 28 days after being diagnosed with COVID-19, including all-cause mortality, requiring invasive mechanical ventilation, or being admitted to the intensive care unit.

SECONDARY OUTCOMES:
all-cause deaths rates | up to 28 days
  The proportion of patients who experienced all-cause mortality within 28 days after being diagnosed with COVID-19.
rehospitalization event rates | up to 28 days
  The proportion of patients who experienced a rehospitalization event within 28 days after being diagnosed with COVID-19
COVID-19 repositive event rates | up to 28 days
  The proportion of patients who experienced a COVID-19 repositive event within 28 days after being diagnosed with COVID-19
adverse drug reaction event | up to 28 days
  The proportion of patients who experienced any adverse drug reaction events within 28 days after being diagnosed with COVID-19.
thromboembolic event rates | up to 28 days
  The proportion of patients who experienced thromboembolic events, including deep vein thrombosis, pulmonary embolism, stroke, and myocardial infarction, within 28 days after being diagnosed with COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Zhang, PhD, Principal Investigator — Beijing Chao Yang Hospital; Zhuoling An, PhD, Principal Investigator — Beijing Chao Yang Hospital; Chaohui Tong, PhD, Principal Investigator — Beijing Chao Yang Hospital

IPD SHARING:
Plan to Share IPD: No